CLINICAL TRIAL: NCT01577953
Title: Phase-Ib Study in Male Patients With Stable Allergic Asthma With Airway Hyperresponsiveness to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Inhaled Single Doses of SB010, a Human GATA-3-specific DNAzyme Solution for Nebulisation - A Randomised, Double-blind, Placebo-controlled, Parallel-group (Per Dose Level) Dose-escalation Study in Asthmatic Patients
Brief Title: Safety, Tolerability, and Pharmacokinetics After a Single Dose of Orally Inhaled DNAzyme Solution for Nebulisation in Male Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sterna Biologicals GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB010/03/2011; 2011-006112-31 (EudraCT Number)
Record Dates: First submitted 2012-04-11; First posted 2012-04-16 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Antisense oligonucleotide; Asthma; Patients with asthma; Phase 1b; Transcription factor GATA-3; Oral inhalation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB010 (Experimental): The drug SB010 is administered in phosphate-buffered saline solution, inhaled via a controlled breathing system over a 5 to 10 min.
  Interventions: Drug: SB010
- Placebo (Placebo Comparator): The placebo (phosphate-buffered saline) is administered as a solution inhaled via a controlled breathing system over a 5 to 10 min.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SB010 — Three consecutive ascending dose groups (A, B, and C) are planned, with a total of 24 patients with asthma. Each dose group will consist of 8 patients (n=6 receiving active drug and n=2 receiving placebo). Each patient will participate in one dose group only.
  Dose escalation to the second and third dose level will occur after satisfactory review of safety and tolerability and after review of the pharmacokinetic data (exposure control, up to 4 hours after administration) of the preceding dose group by the Safety Board.
  Dose levels:
  Dose group A: 5 mg hgd40 in 2 mL solution (concentration: 2.5 mg/mL); Dose group B: 10 mg hgd40 in 2 mL solution (concentration: 5.0 mg/mL); Dose group C: 20 mg hgd40 in 2 mL solution (concentration: 10.0 mg/mL).
  Other Names: The active drug substance of SB010 is hgd40.
  Arms: SB010
Drug: Placebo — Three consecutive ascending dose groups (A, B, and C) are planned, with a total of 24 patients with asthma. Each dose group will consist of 8 patients (n=6 receiving active drug and n=2 receiving placebo). Each patient will participate in one dose group only.
  Dose escalation to the second and third dose level will occur after satisfactory review of safety and tolerability and after review of the pharmacokinetic data (exposure control, up to 4 hours after administration) of the preceding dose group by the Safety Board.
  Arms: Placebo

SUMMARY:
Asthma is a chronic inflammatory bronchial disorder with three distinct components: airway hyper-responsiveness (respiratory hypersensitivity), airway inflammation, and intermittent airway obstruction. One of the characteristics of the disease is an inflammatory reaction of the immune system caused by cytokine production. A substantial number of asthma patients do not satisfactorily respond to steroid therapy and consequently have an unmet medical need for novel targeted therapies with improved specificity, tolerability, and compliance.

Novel therapeutic strategies for the treatment of chronic inflammatory diseases by targeting early disease-causing mechanisms are a promising approach for the treatment of asthma. The transcription factor GATA-3 plays a key role in mediating the asthmatic immune response and has been shown to be necessary and sufficient for the production of cytokines interleukin (IL)-4, IL-5, and IL-13. The active drug substance of the investigational medicinal product SB010 is hgd40. SB010 belongs to a new class of antisense oligonucleotide therapeutics, the 10-23 DNA (deoxyribonucleic acid)zymes (antisense oligonucleotide).

DNAzymes are catalytically active nucleic acids that cleave complementary RNA (ribonucleic acid) molecules. By cleaving GATA-3 mRNA, hgd40 reduces specific cytokine production and thereby reduces key features of allergic airway inflammation. DNAzymes are generated completely by chemical synthesis and can be produced under Good Manufacturing Practice (GMP) controlled conditions. The DNAzymes are not biological drugs, i.e. they are not generated by use of any living organism including cell culture or bacteria. The molecules are highly water-soluble and will be applied as solution directly in their synthesized form.

The current study will evaluate the safety and tolerability of increasing single doses of inhaled SB010 in male patients with asthma who have airway hyperresponsiveness(demonstrated by methacholine bronchial challenge test).

ELIGIBILITY:
Inclusion Criteria:

* Adult male Caucasian patients aged 18-45 years (both included).
* Clinical diagnosis of mild to moderate, stable, persistent or intermittent asthma (according to GINA guidelines revised version 2010) for at least 6 months prior to screening.
* Positive skin reactivity at screening or within the last 12 months to at least one allergen out of a variety of seasonal or non-seasonal specific allergens (e.g. pollen, animal epithelia, dust mite).
* Patients not on concomitant treatments, except for short-acting beta-agonists and inhaled and topical corticosteroids on a stable dose, or able to change current asthma therapy, to discontinue prescribed anticholinergics, leukotriene receptor inhibitors, and long-acting beta 2-agonists after signature of informed consent as per required washout periods.
* Screening forced expiratory volume (FEV1) value of >60% of the predicted normal value after a washout of at least 8 hours for short-acting beta 2-agonists, and 72 hours for long-acting beta 2-agonists, whatever is applicable. Predicted normal values to be used for calculation purposes are to be based on European Community for Steel and Coal predicted values.
* Patients must demonstrate a PC 20 response to methacholine concentrations of ≤4 mg/mL at screening. (PC 20 = Concentration of the agonist in the inhaled substance leading to a fall in FEV1 of 20%).
* Pre-dose FEV1 value not below 20% of the reference absolute FEV1 value measured at screening [i.e. 0.8 x FEV1 (screening) ≥FEV1 pre-dose].
* Patient has been informed both verbally and in writing about the objectives of the clinical trial, the methods, the anticipated benefits and potential risks and the discomfort to which he may be exposed, and has given written consent to participation in the trial prior to trial start and any trial-related procedure.
* Except for asthma or atopic diseases like allergic rhinitis or atopic dermatitis assessed as healthy based on a screening examination including medical history, physical examination, vital signs, ECG assessment, pulmonary function testing, and clinical laboratory results.
* Body weight according to a Body Mass Index ≥18.0 and ≤29.0 kg/m², and a body weight ≥60 and ≤90 kg.
* Non-smokers or ex-smokers who had stopped smoking for at least 5 years prior to start of the clinical study. No history of smoking more than 10 pack-years.
* Ability to inhale in an appropriate manner (patients will be trained to inhale from the AKITA2 APIXNEB® device with a placebo medication at the screening visit).
* The patient must agree:

  * to use two methods of contraception in combination with his female partner, if she is of childbearing potential; this combination of contraceptive methods must be used from screening until at least 6 months after the last dose of Investigational Medicinal Product. At least one of the contraception methods must be a barrier contraception method. Contraceptive methods allowed include the following: condoms, diaphragm in combination with a spermicide, intrauterine device as well as for female partners oral contraception, contraception implants, OR
  * not to be sexually active at screening and accept using double-barrier contraception should he become sexually active during or within 6 months after the last dose of Investigational Medicinal Product, OR
  * to have been surgically sterilized prior to screening and accept to use a barrier method of contraception as well, OR
  * to have a partner who is post-menopausal and has had her last natural menstruation at least 24 months prior to screening, OR
  * to have a partner who has had a hysterectomy prior to screening, OR
  * to have a partner who has been surgically sterilized prior to screening

Exclusion Criteria:

* Presence of clinically significant diseases other than asthma or atopic diseases (cardiovascular, renal, hepatic, gastrointestinal, hematological, neurological, genitourinary, autoimmune, endocrine, metabolic, etc), which, in the opinion of the investigator, may either put the patient at risk because of participation in the trial, or diseases which may influence the results of the study or the patient's ability to take part in it.
* Presence of relevant pulmonary diseases or history of thoracic surgery, such as:

  * Known active tuberculosis
  * Non-small cell lung cancer
  * Pulmonary arterial hypertension
  * History of interstitial lung or pulmonary thromboembolic disease
  * Pulmonary resection during the past 12 months
  * History of allergic asthma
  * History of bronchiectasis secondary to respiratory diseases (e.g., cystic fibrosis, Kartagener's syndrome, etc.)
  * History of chronic bronchitis, emphysema, allergic bronchopulmonary aspergillosis or respiratory infection within the 4 preceding weeks of the first morning IMP administration
* Any absolute or relative contraindications for methacholine challenge: e.g., severe or moderate airflow limitation (FEV1 <60% predicted or <1.5 L), heart attack or stroke in the last 3 months, uncontrolled hypertension, known aortic aneurysm, current use of cholinesterase inhibitor medication.
* Hospitalisation or emergency room treatment for acute asthma in the 3 months prior to screening, between screening and the start of the treatment period.
* Intubation (ever) or hospitalisation for longer than 24 hours for the management of an asthma exacerbation within the preceding 3 months of the screening visit.
* History of allergic reactions to any active or inactive ingredients of the nebuliser solution.
* ECG abnormalities of clinical relevance (e.g., QTc according to Bazett's >440 ms, PR ≥210 ms; or QRS ≥120 ms).
* Patients with a resting heart rate <45 bpm and >90 bpm, systolic blood pressure <100 mmHg and >140 mmHg, diastolic blood pressure <60 mmHg and >90 mmHg.
* Proneness to orthostatic dysregulation, fainting, or blackouts.
* History or presence of any malignancy except for basalioma.
* Clinically relevant abnormalities in clinical chemical, haematological or in any other laboratory variables.
* Chronic or clinically relevant acute infections.
* Positive results in any of the following virology tests: Hepatitis B surface antigen, Hepatitis B core antibodies, Hepatitis C antibodies, human immunodeficiency virus (HIV)-1, and HIV -2 antibodies.
* Positive drug screen.
* History of previous administration of SB010 or any other registered or investigational oligonucleotide-based drug.
* History or presence of alcohol or drug abuse.
* Treatment with any known enzyme inducing or inhibiting agents (St. John's Wort, barbiturates, phenothiazines, cimetidine, ketoconazole etc.) within 30 days before administration of IMP or during the trial.
* Use of any medication (including over-the-counter medication such as herbal products) except allowed concomitant medication within 2 weeks (for biologics: 6 months) before administration of IMP or within <10 times the elimination half-life of the respective drug, or the duration of the pharmacodynamic effect, whatever is longer, or anticipated concomitant medication during the treatment period.
* Consumption of any enzyme inducing or inhibiting aliments and beverages (e.g., broccoli, Brussels sprout, star fruit, etc.) within 14 days prior to administration of IMP or during the trial.
* Consumption of any caffeine- or theophylline-containing product as well as grapefruit and grapefruit-containing products 12 h before administration of IMP.
* Vegetarian diet or other peculiar dietary habits which would preclude the patient's acceptance of standardised meals.
* Surgery of the gastrointestinal tract except for appendectomy or herniotomy.
* Planned donation of germ cells, blood, organs, bone marrow during the course of the trial or within 6 months thereafter.
* Participation in another clinical trial with an investigational drug or device within the last 3 months. For biologics, the minimum exclusion period is at least 6 months or the time of duration of the pharmacodynamic effect or 10 times the half-life of the respective drug whatever is longer before inclusion in this trial.
* Blood donation within the last 30 days before screening.
* Lack of ability or willingness to give informed consent.
* Anticipated non-availability for trial visits/procedures.
* Anticipated lack of willingness or inability to cooperate adequately.
* Vulnerable patients (e.g., persons kept in detention).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Limiting dose of inhaled ascending single dose of SB010. | up to Day 60±4; maximum of 92 days for a particular patient.
  Safety will be monitored as adverse events, vital signs, clinical chemistry, haematology, coagulation, urinalysis, electrocardiogram, pulmonary function testing (serial spirometric measurements), body temperature, overall tolerability. These will be monitored during the study period Days 1 to 4; at the follow up visit Day 12±2; during a follow-up phone call Day 30±3; at the end of study Day 60±4. The maximum duration will be 92 days for a particular patient.

SECONDARY OUTCOMES:
Number of participants with any dose-limiting adverse effects. | during the study period Days 1 to 4; at the follow up visit Day 12±2; during a follow-up phone call Day 30±3; at the end of study Day 60±4; maximum of 92 days for a particular patient.
  Safety will be monitored as adverse events, vital signs, clinical chemistry, haematology, coagulation, urinalysis, electrocardiogram, pulmonary function testing (serial spirometric measurements), body temperature, overall tolerability.
Single-dose plasma concentration of hgd40 over time after inhalation of SB010. | during study period Days 1 to 4.
  The following pharmacokinetic parameters will be determined in plasma samples over 4 days: Area under the plasma concentration-time curve zero to infinity; Area under the plasma concentration-time curve (dose adjusted); Area under the concentration-time curve until the last sampling time; Concentration maximum; Concentration maximum (dose adjusted); Time of maximum concentration; Apparent terminal elimination half-life.
Systemic activity of biomarkers. | at screening Day -28 to -2; during study period Day 1 to 4; at follow up visit day 12±2; at end of study Day 60±4.
  The following biomarkers will be determined in serum (exploratory evaluation): IL-4, IL-5, IL-10, IL-13, IFN-gamma (using validated multiplex immune assay system), and tryptase (using enzyme-linked immunoassay).
  IL=Interleukin; IFN=Interferon.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, Prof. Dr., Principal Investigator — Clinical Airway Research Fraunhofer Institute for Toxicology and Experimental Medicine (ITEM), Hannover, Germany
Locations (1):
- Clinical Airway Research Fraunhofer Institute for Toxicology and Experimental Medicine (ITEM), Hanover, Germany